CLINICAL TRIAL: NCT00942227
Title: The Value of Traction in Treatment of Lumbar Radiculopathy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other); 59th Medical Wing (U.S. Federal Agency); Empi, A DJO Company (Industry)
Responsible Party: Principal Investigator, Julie Fritz, Clinical Outcomes Research Scientist, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1008586
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Sciatica; Radiculopathy; Spinal Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Intervertebral Disk Displacement
Keywords: Sciatica; Radiculopathy; Physical therapy modalities; Rehabilitation
MeSH Terms: conditions — Sciatica; Radiculopathy; Spinal Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extension oriented treatment approach (Active Comparator): Extension exercises. Subjects are instructed in a progression of extension oriented movements for the lumbar spine. Manual therapy may be added to further increase extension movement and/or reduction of symptoms.
  Interventions: Other: Physical therapy rehabilitation
- Mechanical traction plus extension-oriented treatment (Experimental): Mechanical lumbar traction will be utilized in addition to extension oriented exercises. Subjects are also instructed in a progression of extension oriented movements for the lumbar spine. Manual therapy may be added to increase extension movement and/or reduce radicular symptoms.
  Interventions: Other: Physical therapy rehabilitation

INTERVENTIONS:
Other: Physical therapy rehabilitation — Extension oriented exercises. Subjects will be instructed in a progression of extension oriented exercises for the lumbar spine
  Other Names: McKenzie exercises; Directional preference; Specific exercise
  Arms: Extension oriented treatment approach
Other: Physical therapy rehabilitation — Mechanical lumbar traction will be applied with subjects in prone utilizing 40-60% of subject's body weight to create a distraction force in the lumbar spine. Following traction, subjects will be instructed in a progression of extension oriented exercises and manual therapy to increase extension as described for the comparator group.
  Other Names: Saunders 3D Active Trac
  Arms: Mechanical traction plus extension-oriented treatment

SUMMARY:
The purpose of this study is to determine the effectiveness of adding mechanical traction to standard physical therapy treatments for patients with low back pain.

DETAILED DESCRIPTION:
Despite the opinions of clinical experts that patients who might benefit from traction may represent distinct sub-groups of patients, most studies have not attempted to narrow their inclusion criteria beyond loose definitions of 'acute' or 'chronic' symptoms. While these studies seem to indicate that traction interventions will be of little benefit when administered to large groups of patients without a prior attempt to select which patients are most likely to benefit, they are not sufficient to preclude the possibility that a subgroup of patients may benefit substantially from the intervention. Recent preliminary studies suggest a there exists a subgroup of patients with LBP that is likely to benefit from traction.

The two primary aims of this study are:

1. Determine the validity of the previously-identified prediction criteria to identify patients highly likely to benefit from the addition of traction to a standard physical therapy intervention.
2. Compare the overall effectiveness of addition of a traction component to a standard physical therapy intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of pain and/or paresthesia in the lumbar spine with a distribution of symptoms that has extended distal to the gluteal fold on at least one lower extremity within the past 24 hours based on the patient's self-report.
* Oswestry disability score of at least 20%
* Age at least 18 years and less than 60 years
* At least one of the following signs of nerve root compression:

  1. Positive ipsilateral or contralateral straight leg raise test (reproduction of leg symptoms with straight leg raise < 70 degrees)
  2. Sensory deficit to pinprick on the ipsilateral lower extremity
  3. Diminished strength of a myotome (hip flexion, knee extension, ankle dorsiflexion, great toe extension, or ankle eversion) of the ipsilateral lower extremity
  4. Diminished lower extremity reflex (Quadriceps or Achilles) of the symptomatic lower extremity

Exclusion Criteria:

* Red flags noted in the patient's general medical screening questionnaire (i.e., tumor, metabolic diseases, RA, osteoporosis, spinal compression fracture, prolonged history of steroid use, etc.)
* Evidence of central nervous system involvement, to include symptoms of cauda equina syndrome (i.e., loss of bowel/bladder control or saddle region paresthesia) or the presence of pathological reflexes (i.e., positive Babinski)
* Patient reports the complete absence of low back and leg symptoms when seated
* Recent surgery (< 6 months) to the lumbar spine or buttocks, or any fusion surgery of the lumbar spine or pelvis
* Recent (< 2 weeks) epidural steroid injection for low back and/or leg pain
* Current pregnancy
* Inability to comply with the treatment schedule

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | Baseline, 6 weeks, 6 months, 1year

SECONDARY OUTCOMES:
Global Rating of Change | Baseline, 6 weeks, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Fritz, PhD, Principal Investigator — Intermountain Healthcare; University of Utah
Locations (1):
- Intermountain Healthcare, Rehab Agency, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Thackeray A, Fritz JM, Childs JD, Brennan GP. The Effectiveness of Mechanical Traction Among Subgroups of Patients With Low Back Pain and Leg Pain: A Randomized Trial. J Orthop Sports Phys Ther. 2016 Mar;46(3):144-54. doi: 10.2519/jospt.2016.6238. Epub 2016 Jan 26. PMID 26813755
- [Derived] Fritz JM, Thackeray A, Childs JD, Brennan GP. A randomized clinical trial of the effectiveness of mechanical traction for sub-groups of patients with low back pain: study methods and rationale. BMC Musculoskelet Disord. 2010 Apr 30;11:81. doi: 10.1186/1471-2474-11-81. PMID 20433733